CLINICAL TRIAL: NCT02932930
Title: Ultrasound Guided Quadratus Lumborum Block for Postoperative Pain in Abdominoplasty: A Randomized Controlled Study
Brief Title: Ultrasound Guided Quadratus Lumborum Block for Postoperative Pain in Abdominoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, MD, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USJ-02
Record Dates: First submitted 2016-10-10; First posted 2016-10-13 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Pain
Keywords: QLB; Abdominoplasty; Quadratus lumborum block
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- QLB group (Active Comparator): Patients will receive at the beginning of the surgery 0.2 ml/kg of 0.2% ropivacaine bilaterally.
  Procedure: Quadratus Lumborum Block type II, local anesthetic injection on the posterior border of the quadratus lumborum muscle Drug: Ropivacaine, 0.2 ml/kg of 0.2% ropivacaine
  Interventions: Procedure: QLB bloc; Drug: 0.2% Ropivacaine
- Control group (Placebo Comparator): Patients will receive at the beginning of the surgery 0.2 ml/kg of 0.9% normal saline bilaterally.
  Procedure: Quadratus Lumborum Block type II, local anesthetic injection on the posterior border of the quadratus lumborum muscle Drug: Normal saline, 0.2 ml/kg of 0.9 % normal saline
  Interventions: Procedure: QLB bloc; Drug: 0.9% normal saline

INTERVENTIONS:
Procedure: QLB bloc
Drug: 0.2% Ropivacaine — 0,2ml/kg of 0,2% ropivacaine
  Arms: QLB group
Drug: 0.9% normal saline — 0,2ml/kg of 0.9% normal saline
  Arms: Control group

SUMMARY:
The original concept of a quadratus lumborum block (QLB) indicated for analgesia after abdominal surgery was first described by Blanco in 2007. Also referred to as a posterior transversus abdominis plane (TAP) block, the QLB consists in deposition of local anesthetic on either the posterior or the anterolateral border of the quadratus lumborum muscle. TAP blocks have already been proved effective in urologic, abdominal, and gynecologic procedures by blocking the sensory nerve supply to the anterior abdominal wall thus reducing the amount of postoperative analgesic medication. The main advantages of QLB compared to the TAP block is a wider sensory block area and a longer duration of analgesia. This is due to the extension of local anesthetic agents beyond the TAP plane to the thoracic paravertebral space(4).

Previous reports have shown that QLB is effective in providing pain relief after various abdominal operations. However, there are no published reports on QLB for postoperative pain after abdominoplasty. This prospective, randomized, double-blinded, controlled study aims to evaluate the analgesic efficacy, opioids consumption and quality of recovery of QLB in patients undergoing abdominoplasty. Patients scheduled to have abdominoplasty will be randomized to receive bilateral QLB with either ropivacaine 0.2% or normal saline. Post-operative cumulative analgesic medication consumption, pain severity at rest and on movement, as well as quality of recovery will be evaluated and compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Standard abdominoplasty procedure
2. Written informed consent
3. Age ≥ 18 years
4. Female

Exclusion Criteria:

1. Patient's refusal
2. Allergies to any study medication
3. Inability to comprehend or participate in scoring scales
4. Deformations that could possibly affect the spread of the local anesthetic in the quadratus lumborum muscle plane
5. Quadratus lumborum muscle plane not seen in ultrasound examination
6. Coagulopathy or on anticoagulants

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption | up to 48 hour
  Cumulative morphine consumption in mg while in the PACU and tramadol dose till 48 hour post operatively.

SECONDARY OUTCOMES:
Time to first tramadol dose | up to 48 hour
  Time to first tramadol dose: time from the discharge to the surgical ward to the first postoperative subcutaneous tramadol dose requested by the patient.
Postoperative pain severity | up to 48 hour
  Postoperative pain severity in Numerical Rating Scale at rest in the first 48 hour after surgery. Ranging from 0 for no pain to 10 for worst pain imaginable. All patients will be assessed postoperatively by a blinded investigator: at 2, 4, 6, 12, 24, 36, and 48 hour postoperatively.
Postoperative dynamic pain severity | up to 48 hour
  Postoperative dynamic pain severity (walking, coughing, deep breathing) in Numerical Rating Scale in the first 48 hour after surgery. Ranging from 0 for no pain to 10 for worst pain imaginable. All patients will be assessed postoperatively by a blinded investigator: at 2, 4, 6, 12, 24, 36, and 48 hour postoperatively.
Nausea or vomiting | up to 48 hour
  Nausea or vomiting up to 48h post operatively (2, 4, 6, 12, 24, 36, and 48 hour postoperatively) using the following four grades scale:
  0 = No nausea; 1 = Mild nausea; 2 = Moderate nausea; 3 = Severe nausea or vomiting
Sedation level | up to 48 hour
  Sedation level up to 48 hour post operatively using the following Ramsay score.
Quality of recovery | up to 48 hour
  Quality of recovery using the self-assessment quality of recovery (QoR) scale to assess the patient's recovery quality
Time to first walk | up to 48 hour
  Time to first walk

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu De France, Beirut, Aschrafieh, Lebanon

REFERENCES:
- [Background] El-Boghdadly K, Elsharkawy H, Short A, Chin KJ. Quadratus Lumborum Block Nomenclature and Anatomical Considerations. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):548-9. doi: 10.1097/AAP.0000000000000411. No abstract available. PMID 27315184
- [Background] Hockett MM, Hembrador S, Lee A. Continuous Quadratus Lumborum Block for Postoperative Pain in Total Hip Arthroplasty: A Case Report. A A Case Rep. 2016 Sep 15;7(6):129-31. doi: 10.1213/XAA.0000000000000363. PMID 27513972
- [Background] Sforza M, Andjelkov K, Zaccheddu R, Nagi H, Colic M. Transversus abdominis plane block anesthesia in abdominoplasties. Plast Reconstr Surg. 2011 Aug;128(2):529-535. doi: 10.1097/PRS.0b013e31821e6f51. PMID 21788846
- [Background] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Background] Baidya DK, Maitra S, Arora MK, Agarwal A. Quadratus lumborum block: an effective method of perioperative analgesia in children undergoing pyeloplasty. J Clin Anesth. 2015 Dec;27(8):694-6. doi: 10.1016/j.jclinane.2015.05.006. Epub 2015 Jul 11. No abstract available. PMID 26174113
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Chakraborty A, Goswami J, Patro V. Ultrasound-guided continuous quadratus lumborum block for postoperative analgesia in a pediatric patient. A A Case Rep. 2015 Feb 1;4(3):34-6. doi: 10.1213/XAA.0000000000000090. PMID 25642956